CLINICAL TRIAL: NCT02827058
Title: The Influence of Needle Diameter on Needle Failures and Post Dural Puncture Headache in Relation to Cesarean Section and Vaginal Delivery; a Prospective, Randomised Trial
Brief Title: The Influence of Needle Diameter on Post Dural Puncture Headache
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: due to difficulties recruiting patients and therefore too slow progress
Sponsor: Helse Nord-Trøndelag HF (Other)
Collaborators: Sykehuset Ostfold (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2016/140
Record Dates: First submitted 2016-07-06; First posted 2016-07-11 (Estimated); Last update posted 2020-04-24 (Actual); Status verified 2020-04

CONDITIONS: Post-Dural Puncture Headache
Keywords: Delivery, obstetric; Analgesia, Epidural; Injections, Epidural; Needles; Cesarean Section
MeSH Terms: conditions — Post-Dural Puncture Headache; Agnosia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- G25 pencil point needle (Experimental): healthy pregnant women who at (vaginal or cesarean section) delivery get spinal anesthesia administered with use of a 25 gauge pencil point needle
  Interventions: Device: G25 pencil point needle
- G27 pencil point needle (Active Comparator): healthy pregnant women who at (vaginal or cesarean section) delivery get spinal anesthesia administered with use of a 27 gauge pencil point needle
  Interventions: Device: G27 pencil point needle

INTERVENTIONS:
Device: G25 pencil point needle
  Arms: G25 pencil point needle
Device: G27 pencil point needle
  Arms: G27 pencil point needle

SUMMARY:
The purpose of this study is to determine whether injection needle pen point type 'PP Gauge 25' should be recommended as a primary choice of needle (in stead of 'PP Gauge 27') for healthy pregnant women who at delivery (vaginal or cesarean section) get spinal anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* healthy
* pregnant
* spinal anesthesia at delivery (vaginal delivery or cesarean section emergency grade 2-4)
* informed consent

Exclusion Criteria:

* chronic headache
* (attempt to) epidural anesthesia

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 65 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2018-05-01 (Actual); Study Completion 2018-05-01 (Actual)

PRIMARY OUTCOMES:
number of attempts until successful injection | 0 (injection time before delivery)

SECONDARY OUTCOMES:
incidence of post dural puncture headache | 48 hrs

CONTACTS AND LOCATIONS:
Overall Officials: Jan Sverre Vamnes, md, Study Director — Østvold Hospital
Locations (3):
- Norway (3):
  - Østfold Hospital, Fredrikstad
  - Fredrikstad
  - Levanger Hospital, Levanger

IPD SHARING:
Plan to Share IPD: Undecided